CLINICAL TRIAL: NCT00182819
Title: Primary Chemotherapy With Temozolomide Versus Radiotherapy in Patients With Low Grade Gliomas After Stratification for Genetic 1p Loss: A Phase III Study
Brief Title: Radiation Therapy or Temozolomide in Treating Patients With Gliomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: NCIC Clinical Trials Group (Network); British Medical Research Council (Other Government); Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-22033-26033; 2004-002714-11 (EudraCT Number); CAN-NCIC-CE5; TROG 06.01; MRC-BR13
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult oligodendroglioma; adult diffuse astrocytoma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma; Glioma | interventions — Temozolomide; Radiotherapy

ARMS (2):
- radiotherapy (Other): Radiotherapy (control arm), 50.4 Gy, standard fractionation (28 x 1.8 Gy), conformal techniques
  Interventions: Radiation: radiation therapy
- Temozolomide (Experimental): Temozolomide 75 mg/m2 daily x 21 days, q 28 days until progression or for max. 12 cycles (experimental arm)
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — Temozolomide 75 mg/m2 daily x 21 days, q 28 days until progression or for max. 12 cycles
  Arms: Temozolomide
Radiation: radiation therapy — 50.4 Gy, standard fractionation (28 x 1.8 Gy), conformal techniques
  Arms: radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether radiation therapy is more effective than temozolomide in treating gliomas.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared to temozolomide in treating patients with gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of patients with low-grade gliomas treated with radiotherapy vs temozolomide.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Determine whether the incidence of late toxicity can be decreased in patients who are randomized to receive temozolomide.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to participating center, chromosome 1p status (deleted vs normal vs undeterminable), contrast enhancement on MRI (yes vs no), age (< 40 years vs ≥ 40 years), and WHO performance status (0 or 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily, 5 days a week, for a total of 28 fractions (i.e., 5½ weeks).
* Arm II: Patients receive oral temozolomide once daily on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 3 months until disease progression.

After completion of study treatment, patients are followed every 6 months for survival.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A minimum of 699 patients (a total of 466 randomized [233 per treatment arm]) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low-grade glioma, including any of the following types:

  * Astrocytoma (gemistocytic, fibrillary, or protoplasmatic)
  * Oligoastrocytoma
  * Oligodendroglioma
* WHO grade II disease
* Supratentorial tumor location only
* RTOG neurological function 0-3
* Not a candidate for surgical treatment alone
* Requires treatment, as determined by ≥ 1 of the following criteria:

  * Age ≥ 40 years
  * Radiologically-proven progressive lesion
  * New or worsening neurological symptoms other than seizures only (e.g., focal deficits, signs of increased intracranial pressure, or mental deficits)
  * Intractable seizures, defined by both of the following criteria:

    * Experiences persistent seizures that interfere with everyday life activities except driving a car
    * Failed 3 anti-epileptic drug regimens, including ≥ 1 combination regimen
* Tumor material (paraffin-embedded) or histopathologic slides available

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* No chronic hepatitis B or C infection
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No known HIV positivity
* No other serious medical condition
* No other prior or concurrent malignancy except surgically cured carcinoma in situ of the cervix or nonmelanoma skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study participation
* No medical condition that would preclude receiving oral medication (e.g., frequent vomiting or partial bowel obstruction)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent growth factors for elevating absolute neutrophil counts for the purpose of temozolomide administration
* No concurrent epoetin alfa
* No concurrent immunotherapy or biologic therapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy, including adjuvant chemotherapy for patients randomized to undergo radiotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the brain
* No concurrent integrated boost with intensity-modulated radiotherapy

Surgery

* Recovered from prior surgery
* No concurrent surgical tumor debulking

Other

* No prior randomization to this study
* No other concurrent investigational drugs
* No concurrent regular use of agents known to be radiosensitizers or radioprotectors (e.g., cyclooxygenase-2 inhibitors, thalidomide, or amifostine) during study radiotherapy

  * Occasional use of nonsteroidal anti-inflammatory drugs for pain allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2005-07; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Quality of life as measured by QLQ-C30 v3.0 and EORTC BN-20 | every 3 months until progression, and then every 6 months until death
Mini-Mental State Examination | every 3 months until progression, and then every 6 months until death
Adverse events as measured by CTCAE v3.0 | As indicated in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Baumert, MD, PhD, Study Chair — Maastricht University Medical Center; Roger Stupp, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (89):
- Australia (12):
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin and Repatriation Medical Centre, Heidelberg West, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital - Nedlands, Nedlands, Western Australia
  - Liverpool Hospital, Liverpool
- Medical University Vienna - General Hospital AKH, Vienna, Austria
- Belgium (3):
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Canada (12):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Mcgill University Health Centre - Gerald Bronfman Centre - Dept Of Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - BC Cancer Agency, Vancouver
- National Cancer Institute of Egypt, Cairo, Egypt
- France (10):
  - CHU de Bordeaux - Groupe Hospitalier Saint-André - Hopital Saint-Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - CHU de la Timone, Marseille
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (4):
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetskliniken Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen, Tübingen
- National Institute Of Neurosurgery, Budapest, Hungary
- Rambam Health Care Campus, Oncology Institute, Haifa, Israel
- Italy (4):
  - Ospedale Bellaria, Bologna
  - Ospedale San Raffaele, Milan
  - Istituto Regina Elena / Istituti Fisioterapici Ospitalieri, Roma
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
- Centre Francois Baclesse, Esch / Alzette, Luxembourg
- Netherlands (8):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastro Clinic - Maastricht Radiation Oncology, Maastricht
  - Radboud University Medical Center Nijmegen, Nijmegen
  - Erasmus MC Cancer Institute - location Daniel den Hoed, Rotterdam
  - Medisch Centrum Haaglanden - Westeinde, The Hague
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Canterbury Health Laboratories, Christchurch, New Zealand
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, SA, Lisbon, Portugal
- National University of Singapore, Singapore, Singapore
- Spain (6):
  - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona - (Barcelona)
  - Hospital General Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico Universitario de Barcelona, Barcelona
  - ICO Girona - Hospital Doctor Josep Trueta (Institut Catala D'Oncologia), Girona
  - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), L'Hospitalet de Llobregat
- Sweden (4):
  - University Hospital of Linkoping, Linköping
  - Skane University Hospital, Lund
  - Umea Universitet, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (3):
  - Oncology Institute of Southern Switzerland - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (15):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol, Avon
  - Clatterbridge Centre for Oncology, Bebington, Wirral, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - University College Hospital, London, England
  - Royal Marsden - London, London, England
  - Christie Hospital, Manchester, England
  - James Cook University Hospital, Middlesbrough, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Marsden - Surrey, Sutton, England
  - Gloucestershire Hospital NHS Foundation Trust - Cheltenham General Hospital, Cheltenham
  - Western General Hospital, Edinburgh
  - Royal Free Hospital, London
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford
  - Lancashire Teaching Hospitals NHS Foundation Trust - Royal Preston Hospital, Preston

REFERENCES:
- [Background] Musat E, Roelofs E, Bar-Deroma R, Fenton P, Gulyban A, Collette L, Stupp R, Weber DC, Bernard Davis J, Aird E, Baumert BG. Dummy run and conformity indices in the ongoing EORTC low-grade glioma trial 22033-26033: First evaluation of quality of radiotherapy planning. Radiother Oncol. 2010 May;95(2):218-24. doi: 10.1016/j.radonc.2010.03.005. Epub 2010 Apr 6. PMID 20378192
- [Background] Fairchild A, Weber DC, Bar-Deroma R, Gulyban A, Fenton PA, Stupp R, Baumert BG. Quality assurance in the EORTC 22033-26033/CE5 phase III randomized trial for low grade glioma: the digital individual case review. Radiother Oncol. 2012 Jun;103(3):287-92. doi: 10.1016/j.radonc.2012.04.002. Epub 2012 May 3. PMID 22560713
- [Derived] Gao Y, Weenink B, van den Bent MJ, Erdem-Eraslan L, Kros JM, Sillevis Smitt P, Hoang-Xuan K, Brandes AA, Vos M, Dhermain F, Enting R, Ryan GF, Chinot O, Ben Hassel M, van Linde ME, Mason WP, Gijtenbeek JMM, Balana C, von Deimling A, Gorlia T, Stupp R, Hegi ME, Baumert BG, French PJ. Expression-based intrinsic glioma subtypes are prognostic in low-grade gliomas of the EORTC22033-26033 clinical trial. Eur J Cancer. 2018 May;94:168-178. doi: 10.1016/j.ejca.2018.02.023. Epub 2018 Mar 20. PMID 29571083
- [Derived] Baumert BG, Hegi ME, van den Bent MJ, von Deimling A, Gorlia T, Hoang-Xuan K, Brandes AA, Kantor G, Taphoorn MJB, Hassel MB, Hartmann C, Ryan G, Capper D, Kros JM, Kurscheid S, Wick W, Enting R, Reni M, Thiessen B, Dhermain F, Bromberg JE, Feuvret L, Reijneveld JC, Chinot O, Gijtenbeek JMM, Rossiter JP, Dif N, Balana C, Bravo-Marques J, Clement PM, Marosi C, Tzuk-Shina T, Nordal RA, Rees J, Lacombe D, Mason WP, Stupp R. Temozolomide chemotherapy versus radiotherapy in high-risk low-grade glioma (EORTC 22033-26033): a randomised, open-label, phase 3 intergroup study. Lancet Oncol. 2016 Nov;17(11):1521-1532. doi: 10.1016/S1470-2045(16)30313-8. Epub 2016 Sep 27. PMID 27686946
- [Derived] Reijneveld JC, Taphoorn MJB, Coens C, Bromberg JEC, Mason WP, Hoang-Xuan K, Ryan G, Hassel MB, Enting RH, Brandes AA, Wick A, Chinot O, Reni M, Kantor G, Thiessen B, Klein M, Verger E, Borchers C, Hau P, Back M, Smits A, Golfinopoulos V, Gorlia T, Bottomley A, Stupp R, Baumert BG. Health-related quality of life in patients with high-risk low-grade glioma (EORTC 22033-26033): a randomised, open-label, phase 3 intergroup study. Lancet Oncol. 2016 Nov;17(11):1533-1542. doi: 10.1016/S1470-2045(16)30305-9. Epub 2016 Sep 27. PMID 27686943